CLINICAL TRIAL: NCT04668170
Title: Identification of Predictive Immune Biomarkers Based on the Understanding of COVID-19 Pathogenesis to Influence Therapeutic Management
Brief Title: Predictive Immune Biomarkers of COVID-19 Pathogenesis to Influence Therapeutic Management
Acronym: IMMUNOMARKCOV
Status: Completed | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/20/0187
Record Dates: First submitted 2020-11-12; First posted 2020-12-16 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: COVID-19
Keywords: SARS-CoV-2; predictive medicine; pathophysiology; immune responses
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- hospitalized patients: very well-defined population of COVID-19 patients with the following outcomes:
  Patients with severe disease requiring on admission ICU management for SARS, Non-severe hospitalized patients with secondary clinical worsening requiring ICU management, Non-severe hospitalized patients without clinical worsening requiring ICU management.
  Interventions: Biological: Blood collection on admission and longitudinally
- healthcare workers: mildly symptomatic patients among healthcare workers attending outpatient dedicated clinics will be recruited
  Interventions: Biological: Blood collection on their first consultation and 10 to 14 days later

INTERVENTIONS:
Biological: Blood collection on admission and longitudinally — Samples already collected on admission (day 0) and longitudinally (day 4, 8 12 and in discharge)
  Groups: hospitalized patients
Biological: Blood collection on their first consultation and 10 to 14 days later — Samples already collected on consultation (D0) and 14 days later
  Groups: healthcare workers

SUMMARY:
Persons infected with Severe Acute Respiratory Syndrome (SARS) SARS-CoV-2 vary in severity from being asymptomatic to having fever, cough, sore throat, general weakness and fatigue and muscular pain and in the most severe cases, severe pneumonia, acute respiratory distress syndrome and sepsis potentially leading to death. Predictive markers of clinical worsening after admission are lacking. COVID-19 immunopathogenesis and relevant therapeutic strategies are still under investigation.

Although viral shedding peaks during the first week of symptoms, reports show that clinical deterioration often coincides with the development of host antiviral immune responses. The inflammatory response to SARS-CoV-2 infection may underpin COVID-19 pathogenesis leading to aberrant and excessive immune responses that may enter the pulmonary circulation in large numbers and play an immune damaging role causing lung functional disability resulting in clinical worsening. Therapeutic strategies using corticosteroids or biotherapies targeting IL-6 may be valuable in some patients. Based on a better understanding of COVID-19 immunopathogenesis, the identification of predictive biomarkers early in the disease process would be of outstanding interest to tailor prompt therapeutic interventions.

On these bases, the present project aims to unravel, using innovative integrated multimodal immunological approaches, immunologic predictive markers by finely characterizing from their admission innate and adaptive immune responses in two well described cohorts of COVID-19 patients that are being collected in Toulouse (COVID-BioToul) and Bordeaux (COLCOV-19 BX).Those two biological cohorts are connected with two clinical cohorts in Toulouse and Bordeaux in order to have a very well defined population of COVID-19 patients and their clinical outcome. In both cohorts, investigators harvest and cryopreserve biological samples, including plasma and peripheral blood mononuclear cells (PBMCs), on admission and longitudinally from patients evolving or not toward severe forms of the disease in Bordeaux and Toulouse University Hospitals and will allow to investigate primary and secondary objectives. Moreover in the two centers, there are also two clinical outpatients cohorts of healthcare workers attending dedicated clinics in the frame of their surveillance medical program, which constitute groups of patients with benign forms of COVID-19.

DETAILED DESCRIPTION:
The primary objective of IMMUNOMARK-COV is to define an applicable immune signature predicting clinical worsening on COVID-19 patient admission in order to help physicians to take informed therapeutic decisions able to modify early the course of the disease.

Secondary objectives are:

* To assess the early dynamics of SARS-CoV-2-specific cellular immunity in patients followed longitudinally
* To assess the dynamics of gd T cells during COVID-19
* Transcriptomic analysis of discrete and functionally major T cell populations
* To assess SARS-CoV-2-specific humoral immunity in patients upon recovery

Identification of early predictive biomarkers of worsening of COVID-19 patients is of paramount importance. This goal is expected to be achieved through the fine analysis of circulating immune effectors, and their dynamics, in categories of patients with very different clinical outcomes.

To date, management of clinical worsening relies mainly on supportive care in ICU, leading to prolonged stay and saturation of facilities. Earlier therapeutic intervention based on identification of robust predictive biomarkers should:

* Help physicians to take therapeutic decisions
* Improve prognosis of patients that suffered from clinical worsening
* Prevent clinical worsening and transfer to ICU
* Improve the burden relying on ICU facilities in a setting of overflow
* Improve the prevention and management of COVID-19 patients to be able to face in a near future several other waves of COVID-19 Furthermore, identification of immune effectors implicated in tissular damages may also help to identify new therapeutic targets.

ELIGIBILITY:
Inclusion Criteria:

For COVID-19 hospitalized patients

* Polymerase chain reaction (PCR) proven SARS-CoV-2 infection
* Participation to Toulouse clinical cohort
* Having signed consent for inclusion in the Toulouse biobanks For COVID-19 healthcare workers attending dedicated clinics
* PCR proven SARS-CoV-2 infection
* Having signed consent for inclusion in the Toulouse biobanks

Exclusion Criteria:

* Pregnancy or breastfeeding
* Participation in another interventional clinical study involving exploratory treatment or blood sampling.

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized or healthy workers for COVID-19
Sampling Method: Non-Probability Sample
Enrollment: 304 (Actual)
Dates: Start 2020-05-05 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2023-05-02 (Actual)

PRIMARY OUTCOMES:
Immune signature on admission : phenotypic profile of blood T-cells | Day 0
  Immune signature will be compared between COVID-19 patients according to their clinical characteristics and outcome, together with SARS-CoV2 viral shedding (known for every patient in the cohort) on samples harvested on admission: a phenotypic profiling of blood T-cells by multicolor FACS analysis (using 30+ color panels analyzed by multiparametric flow cytometry) assessing T cell subsets (classical CD4 or CD8 T-cells as well as unconventional gdT-cells and regulatory T cells) through the expression of a wide range of surface and intracellular markers.
Immune signature on admission : inflammatory cytokines | Day 0
  Immune signature will be compared between COVID-19 patients according to their clinical characteristics and outcome, together with SARS-CoV2 viral shedding (known for every patient in the cohort) on samples harvested on admission: An analysis on plasma samples of concentration of a wide range of inflammatory cytokines such as IFNa, IFNb and IL-6.

SECONDARY OUTCOMES:
Dynamics of cellular immunity: CD4 and CD8 T cells | Day 0, Day 4, Day 8, Day 12, Day 30 (or in discharge)
  On samples harvested longitudinally from patients, analysis of the relative magnitude and dynamic and polyfunctional profile of SARS-CoV-2 specific CD8 and CD4 T cell responses by analyzing the capacity of T cells to produce simultaneously a variety of cytokines such as IFNa, IFNb and IL-6, will be performed.
Dynamics of cellular immunity: gd T cells | Day 0, Day 4, Day 8, Day 12, Day 30 (or in discharge)
  On samples harvested longitudinally from patients, dynamics of gd T cells will be performed.
Dynamics of cellular immunity: T cell transcriptomic analysis | Day 0, Day 4, Day 8, Day 12, Day 30 (or in discharge)
  On samples harvested longitudinally from patients, transcriptomic analysis of different types of T cells will be performed.
Dynamics of cellular immunity: humoral immunity | Day 0, Day 4, Day 8, Day 12, Day 30 (or in discharge)
  On samples harvested longitudinally from patients, humoral immunity will be performed.

CONTACTS AND LOCATIONS:
Overall Officials: Pierre DELOBEL, MD PhD, Principal Investigator — University Hospital, Toulouse
Locations (2):
- France (2):
  - University Hospital Bordeaux, Bordeau
  - University Hospital Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: No